CLINICAL TRIAL: NCT04717557
Title: Hyperbaric Oxygen Therapy to Prevent Complications After Lower Limb Amputation
Brief Title: Hyperbaric Oxygen and Outcome After Below Knee Amputations
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: low enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00093687
Record Dates: First submitted 2021-01-13; First posted 2021-01-22 (Actual); Results first posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Amputation; Postoperative, Sequelae
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Permuted block
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hyperbaric Oxygen Plus Regular Care (Experimental): Hyperbaric oxygen (2 hours at 2 atmospheres absolute) to be administered 1-2 times daily for up to 10 treatments after amputation. Usual care for patients with amputation (dressing changes and treatment of infection) will be administered in parallel.
  Interventions: Drug: Hyperbaric Oxygen
- Regular Care (No Intervention): Usual care for patients with amputation, including dressing changes and treatment of infection.

INTERVENTIONS:
Drug: Hyperbaric Oxygen — Hyperbaric oxygen (HBO2) 1-2 times daily for up to 10 times after amputation
  Other Names: HBO2
  Arms: Hyperbaric Oxygen Plus Regular Care

SUMMARY:
This study is being conducted to assess the utility of hyperbaric oxygen as an adjunctive treatment to reduce postoperative complications. It is hypothesized that HBO2 given in the immediate postoperative period will reduce postoperative complications in patients undergoing below-the-knee amputations. The objective of this study will be to compare treatment and standard care groups, randomly created of eligible patients, to compare their postoperative complications and to assess their postoperative hospital length of stay, 90-day mortality, failure to heal at 4 and 8 week follow-up visits and ability to ambulate with a prosthesis at 6 months post amputation.

DETAILED DESCRIPTION:
This is a clinical study to test the hypothesis that Hyperbaric Oxygen (HBO2) given in the immediate postoperative period for a total of 10 treatments after Below-the-Knee Amputation (BKA) for vascular disease will reduce postoperative complications. Patients scheduled for BKA at Duke University Medical Center will be reviewed for contraindications to HBO2. Patients for whom HBO2 is not contraindicated may choose to be enrolled in the study. Patients enrolled will be randomly assigned to receive treatment or standard postoperative care. Each patient receiving treatment will receive twice daily HBO2 for 2 hours at breathing 100% oxygen at 2 atmospheres absolute (ATA). Patients receiving HBO2 will breathe 100% oxygen via head tent while inside a hyperbaric chamber at Duke University Hospital. The statistical plan for this study will test non-directional hypotheses (two-sided tests). Bonferroni correction will be used to adjust for multiple tests. The main analysis of the primary efficacy hypotheses will include data from all randomized patients in the group to which random assignment is made. Hence, the analysis will be intention to treat. This study will primarily aim to assess whether patients receiving treatment suffer fewer complications, as defined by the Vascular Quality Initiative, vs. patients who receive standard care. The Vascular Quality Initiative (VQI) is a multicenter voluntary reporting system for outcomes related to vascular surgery. The primary outcome of this study, postoperative complications, will be those outcomes meeting the definition set out in the VQI data dictionary, the set of definitions for inclusion in the VQI database. This allows for a standard definition of complications recognized by a majority of US academic medical centers. Secondary outcomes include hospital length of stay, 90-day mortality, failure to heal at 4 and 8 week follow-up visits and ability to ambulate with a prosthesis at 6 months post amputation.

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* Non-traumatic indication for lower limb amputation
* Able to receive hyperbaric oxygen therapy

Exclusion Criteria:

* Unable to consent
* Contraindication to hyperbaric oxygen
* End stage renal disease on dialysis
* Current renal failure as measured by creatinine levels vs baseline change of more than 1 mg/dL and for whom dialysis is expected to be required with the next month
* Calciphylaxis
* Traumatic injuries that are the cause of the amputation
* Cancer being treated by chemotherapy, scheduled to be treated, or being treated or scheduled to be treated by radiation.
* Limb amputation secondary to ischemic complications from other operations
* Second amputation or reoperation on prior amputation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was in hospital.
Groups:
- Hyperbaric Oxygen Plus Regular Care: Hyperbaric oxygen (2 hours at 2 atmospheres absolute) to be administered 1-2 times daily for up to 10 treatments after amputation. Usual care for patients with amputation will be administered in parallel.
  Hyperbaric Oxygen: Hyperbaric oxygen (HBO2) 1-2 times daily for up to 10 times after amputation
- Regular Care: Usual care for patients with amputation.
Period: Overall Study
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Started | 3 | 1
Completed | 0 | 1
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: years] | 52 [31 to 74] | 74 [74 to 74] | 57.5 [31 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mortality During the Inpatient Period
Time Frame: During inpatient stay immediately after amputation, up to 13 days
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 3 | 1
Participants | 1 | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p = 1.0, Chi-squared
Statistical Analysis 2: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p > 0.5, Chi-squared, Corrected — Underpowered due to early termination

2. Primary Outcome: Number of Participants With Re-operation
Description: Unplanned return to the OR (operating room) for a surgical procedure
Time Frame: Up to 90 days after amputation
Population: One participant in the Hyperbaric Oxygen Plus Regular Care arm died following amputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p > 0.5, Chi-squared, Corrected — Underpowered due to early termination

3. Primary Outcome: Number of Participants With Wound Infection
Description: Any wound site infection that was culture positive or required antibiotic treatment
Time Frame: Up to 90 days after amputation
Population: One participant in the Hyperbaric Oxygen Plus Regular Care arm died following amputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p > 0.5, Chi-squared, Corrected — Underpowered due to early termination

4. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay immediately after amputation
Time Frame: up to approximately 30 days
Measure: Mean (Full Range); unit: days
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 3 | 1
days | 5.3 [4 to 7] | 13 [13 to 13]
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p > 0.5, t-test, 2 sided — Underpowered due to early termination

5. Secondary Outcome: Number of Participants With 90-day Mortality
Description: Death within 90 days after amputation
Time Frame: Up to 90 days after amputation
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 3 | 1
Participants | 1 | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Underpowered - no statistically significant difference; Test type: Superiority; p > 0.5, Cochran-Mantel-Haenszel

6. Secondary Outcome: Number of Participants With Complete Healing of Amputation Wound Healing at 4 Weeks Following Surgery
Description: Complete wound healing at 4 weeks after amputation
Time Frame: 4 weeks after amputation
Population: One participant in the Hyperbaric Oxygen Plus Regular Care arm died following amputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p > 0.5, Chi-squared, Corrected — Underpowered due to early termination

7. Secondary Outcome: Number of Participants With Complete Healing of Amputation Wound Healing at 8 Weeks Following Surgery
Description: Complete wound healing at 8 weeks after amputation
Time Frame: 8 weeks after amputation
Population: One participant in the Hyperbaric Oxygen Plus Regular Care arm died following amputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 2 | 1
Participants | 1 | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p > 0.5, Chi-squared, Corrected — Underpowered due to early termination

8. Secondary Outcome: Number of Participants Able to Ambulate With Prosthesis
Description: Ability to ambulate with a prosthesis at 6 months post amputation
Time Frame: 6 months after amputation
Population: One participant in the Hyperbaric Oxygen Plus Regular Care arm died following amputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 2 | 1
Participants | 2 | 0
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p > 0.5, Chi-squared, Corrected — Underpowered due to early termination

9. Other Pre Specified Outcome: Number of Participants With Hospital Readmission
Description: Any readmission to hospital after initial discharge
Time Frame: Up to 90 days after amputation
Population: One participant in the Hyperbaric Oxygen Plus Regular Care arm died following amputation.
Measure: Count of Participants; unit: Participants
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1
Statistical Analysis 1: Comparison: Hyperbaric Oxygen Plus Regular Care vs Regular Care; Test type: Superiority; p > 0.5, Chi-squared, Corrected — Underpowered due to early termination

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Hyperbaric Oxygen Plus Regular Care | Regular Care
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

LIMITATIONS AND CAVEATS:
Due to insufficient recruitment the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-16): https://cdn.clinicaltrials.gov/large-docs/57/NCT04717557/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT04717557/ICF_001.pdf